CLINICAL TRIAL: NCT01822990
Title: Influence of Circulating Anti-beta2-glycoprotein I Antibodies on the Endothelial Function and NO Metabolism in Peripheral Arterial Disease Patients.
Brief Title: Circulating Anti-Beta2-glycoprotein Antibodies and Endothelial Dysfunction
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Joaquin de Haro, M.D., Study director, Hospital Universitario Getafe
Other Study IDs: ABGPINO150613
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Anti-beta2-glycoprotein antibodies; Peripheral arterial disease; Inflammation; Nitric oxide; Endothelial dysfunction
MeSH Terms: conditions — Peripheral Arterial Disease; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Serum samples of all the subjects included.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atherosclerotic patients: Male patients with intermittent claudication.
- Control subjects: healthy male subjects with normal results on vascular examination and no cardiovascular risk factors, who are not in receipt of any pharmacological treatment, matched by age within two years with peripheral arterial disease patients

SUMMARY:
Circulating anti-beta2-glycoprotein antibodies have been associated with coronary artery disease and peripheral arterial disease. This auto-antibodies could activate endothelial cells leading to the expression of leukocyte adhesion molecules and increasing the release of pro-inflammatory cytokines.

On the other hand, endothelial dysfunction of atherosclerotic patients acts as a primary pathogenic event, as it occur before structural changes are evident on angiogram or ultrasound scan. Loss of endothelial normal function causes vasoconstriction, local coagulation alterations and an increase arterial wall proliferation. This situation s been attributed to a reduction in nitric oxide bioactivity, and to an increase oxygen-free radical formation in the context of the pro-inflammatory status found in atherosclerosis.

Hypothesis: Circulating Anti-beta2-glycoprotein I antibodies could be associated with endothelial dysfunction and nitric oxide metabolism disruption en patients with peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Peripheral arterial disease diagnosis
* Intermittent claudication.
* Hemodynamic confirmation of the disease through non-invasive vascular studies.

Exclusion Criteria:

* Autoimmune disease
* Previous revascularization of the ischemic limb.
* Ischemic ulcers
* Previous history of organ transplants.
* Treatment with immunosuppressors

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: Male patients with intermittent claudication due to peripheral arterial disease after haemodynamic confirmation of the disease by Doppler and treadmill exercise testing. No previous history of autoimmune disease.
  Controls: Healthy male subjects with normal results on vascular examination and no cardiovascular risk factors, who were not in receipt of any pharmacological treatment, matched by age within two years with PAD patients.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Circulating anti-beta2-glycoprotein I antibodies | 12 months
  The titer of circulating anti-endothelial cell antibodies directed against beta2-glycoprotein antigens (Circulating ABGPI) could be detected by indirect immunofluorescence using a diagnosis reagent kit and subjects serum.
Flow-mediated arterial dilatation (FMAD) | 12 months
  FMAD is an ultrasound test based on the ability of endothelial cells to detect changes in shear stress and is one of the most effective and reliable indirect methods for estimating endothelial dysfunction. The ultrasound transducer is applied proximal to the antecubital fossa, and a longitudinal image of the brachial artery is obtained. The basal arterial diameter is determined. A blood pressure cuff is then placed distal to the measurement area and inflated to a pressure of 250 mmHg for five minutes. New measurements of the arterial diameter in the final diastolic phase should be obtained, 60 seconds after the cuff is deflated
Nitrite serum levels | 12 months
  Nitrite serum levels reflects the nitric oxide metabolism. Serum nitrite concentration could be measured by colorimetric analysis using the Griess reaction. This is a chemical reaction which uses sulphanilamide and naphthylethylenediamine dihydrochloride under acid conditions (phosphoric acid).The system is capable of detecting nitric oxide in a variety of biological and experimental fluids, like human serum samples.
Highly sensitive C-reactive protein. | 12 months
  Highly sensitive C-reactive protein levels could be measured using a highly sensitive, automated immunoassay with the human serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Varela, MD, Principal Investigator — Hospital Universitario de Getafe; Joaquin De Haro, MD, Study Director — Hospital Universitario de Getafe; Francisco Acin, MD, PhD, Study Director — Hospital Universitario de Getafe
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain